CLINICAL TRIAL: NCT04566055
Title: Assessing AlloSure Dd-cfDNA Monitoring Insights of Renal Allografts With Longitudinal Surveillance
Acronym: ADMIRAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: ADMIRAL
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Plasma from venous blood will be collected and cell-free DNA will be extracted from the plasma for analysis of donor-derived cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Prospective observational cohort
  Interventions: Device: AlloSure

INTERVENTIONS:
Device: AlloSure — Patients will receive donor-derived cell-free DNA testing for surveillance and for-cause.

SUMMARY:
Prospective Observational Multicenter Cohort. External validation of donor derived cell free DNA in Renal Transplantation. Assessing performance of dd-cfDNA as a surveillance tool and its association with clinical outcomes. Outcomes include formation of de-novo DSA, eGFR decline, performance of AlloSure dd-cfDNA in Allograft rejection.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patients

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Renal transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Validation of AlloSure in Allograft rejection | October 2020

SECONDARY OUTCOMES:
Performance of AS with De-Novo DSAs, Performance in subclinical and protocol biopsies vs clinically indicated for cause biopsies, Survival analysis considering AS surveillance | October 2020

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Colorado Hospital, Aurora, Colorado
  - Tampa General Hosptial, Tampa, Florida
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Hermann Hosptial, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided